CLINICAL TRIAL: NCT03702764
Title: Definition: Impact of Coronary Plaque Geometry on Plaque Vulnerability and Their Association With the Risk of Future Cardiovascular Events in Patients With Chest Pain Undergoing Coronary Computed Tomographic Angiography - the GEOMETRY STUDY
Brief Title: Coronary Plaque Geometry and Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: University of Targu Mures, Romania (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0218-GEO
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-07

CONDITIONS: Coronary Stenosis; Acute Coronary Syndrome; Acute Myocardial Infarction; Atherosclerosis; Atheromatous Plaques
Keywords: coronary plaque eccentricity; vulnerable coronary plaque; coronary artery disease; myocardial infarction; coronary computed tomography angiography; major adverse cardiac events
MeSH Terms: conditions — Coronary Stenosis; Acute Coronary Syndrome; Atherosclerosis; Plaque, Atherosclerotic; Coronary Artery Disease; Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- VP-SG 01: Study subjects that present concentric coronary plaques
  Interventions: Diagnostic Test: CCTA
- VP-SG 02: Study subjects that present eccentric coronary plaques
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — 128-multislice CT coronary angiography and complex atherosclerotic plaque analysis, with the use of CT imaging post-processing techniques.

SUMMARY:
The aim of GEOMETRY study is to investigate the correlation between coronary plaque geometric modifications and lesion vulnerability in patients with suspected coronary artery disease referred for cardiac computed tomography angiography (CCTA). Furthermore the study will evaluate the impact of plaque eccentricity and morphology on the rate of major adverse cardiovascular events (MACE) for a 2 years follow-up period.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the leading cause of mortality and morbidity worldwide. Early detection of CAD may reduce the incidence of myocardial infarction by improving primary prevention and providing more effective treatment methods. A step in this direction is identifying the pattern of coronary plaques which are prone to rupture. Coronary computed tomography angiography (CCTA) has emerged recently as a reliable noninvasive tool used in the evaluation of coronary arteries. Some features related to plaque composition and morphology such as low attenuation plaques, spotty calcification, positive remodeling or napkin ring sign, were already identified as vulnerability markers. However the role of lesion geometry on plaque vulnerability was not investigated yet.

This is a prospective, cohort, single-center study which will be carried out in the Center of Advanced Research in Multimodal Cardiac Imaging Cardiomed.

The study will include 1.000 subjects with suspected CAD who are referred to CCTA by the attending physician and in which presence of at least one coronary plaque is confirmed by CCTA.

Plaque burden, composition, and morphology will be assessed for each plaque. Longitudinal and transversal eccentricity will be also assessed in each plaque and in all cases, eccentricity index will be calculated in cross-section plane at the degree of maximum stenosis in order to determine the position of the remaining circulant lumen and to classify the plaque into concentric and eccentric lesion.

The study will be conducted over a period of 3 years, in which patients will be examined at baseline, and will be followed-up for 2 years for occurrence of MACE.

Study objectives:

Primary: to evaluate the association between different patterns of plaque geometry and the risk for major adverse cardiac events MACE (all-cause mortality, cardiovascular death, myocardial infarction, repeated revascularization, repeated hospitalizations for cardiovascular related incidents, cerebrovascular events) during a 2-year follow-up, Secondary: to evaluate the association of plaque eccentricity, plaque vulnerability and plaque progression after 2 years of follow-up

Study Timeline:

* Baseline (day 0)

  * Obtain and document consent from participant on study consent form.
  * Verify inclusion/exclusion criteria.
  * Obtain demographic information, medical history, medication history, alcohol and tobacco use history.
  * Record results of physical examinations and 12-lead ECG.
  * Collect blood specimens.
  * Imaging: 128-multislice CT angiography.
* Visit 1 (month 6)

  * Record results of physical examinations, 12-lead ECG and medical history.
  * MACE assessment
* Visit 2 (month 12)

  * Record results of physical examinations, 12-lead ECG and medical history.
  * MACE assessment
* Visit 3 (month 18)

  * Record results of physical examinations, 12-lead ECG and medical history.
  * MACE assessment
* Final study visit (month 24)

  * Record results of physical examinations, 12-lead ECG and medical history.
  * Repeat CCTA and plaque assessment
  * End-point evaluation.

Study procedures:

* Medical history, clinical examination, laboratory tests;
* 12-lead ECG
* 128-multislice CT coronary angiography with the evaluation of: calcium score, plaque burden, markers for lesion severity (degree of stenosis, lesion length, lumen area and diameter, minimum and maximum plaque thickness); morphological plaque characteristics (plaque related volumes, plaque burden, remodeling indexes); shear stress by computational fluid dynamics; markers of plaque vulnerability (low attenuation plaque, spotty calcification, positive remodeling, napkin ring sign); plaque geometry by eccentricity index, longitudinal and transversal eccentricity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected coronary artery disease (CAD) and pre-test probability of CAD between 15% and 85%, who undergo CCTA, and in whom CCTA has identified presence of at least one coronary plaque
* Ability to provide informed consent
* Age grater then 18 years

Exclusion Criteria:

* Patients with pre-test probability of CAD >85% or <15%
* Electrocardiographic evidence of STEMI
* Presence of pre-existing CAD including prior myocardial infarction
* History of coronary artery revascularization (by percutaneous coronary intervention, stent or bypass graft surgery)
* Atrial fibrillation or other irregular rhythm
* Unwillingness or incapacity to provide informed consent
* Allergy to iodine contrast media
* Inability to tolerate beta-blocker medication
* Renal insufficiency (creatinine greater than 1.5 mg/dL) or renal failure requiring dialysis
* Pregnant women or lactation
* Active malignancy or malignancy within the last 5 year prior to enrolment
* Conditions associated with an estimated life expectancy of under 2 years
* Coronary calcium score >1000

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population includes patients from a single center with suspected coronary artery disease, meeting inclusion and exclusion criteria and undergoing CCTA by physician referral for coronary luminal evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | Month 24
  Incidence of MACE during follow-up

SECONDARY OUTCOMES:
Coronary plaque vulnerability associated to plaque eccentricity | Month 24
  Number of vulnerability markers in eccentric vs concentric plaques

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Mureș County, Romania